CLINICAL TRIAL: NCT01798537
Title: Simplified Selective Digestive Tract Decontamination for the Prevention of ICU Infections in the Setting of High-level Antibiotic Resistance
Brief Title: Simplified Selective Digestive Tract Decontamination for the Prevention of Intensive Care Unit Acquired Infections
Acronym: SDDICU
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 0401-12-RMB CTIL; NIHP Israel (Other: Israel National Institute for Health Policy)
Record Dates: First submitted 2013-02-17; First posted 2013-02-26 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Bacteremia Associated With Intravascular Line; Ventilator Associated Pneumonia; Bacteremia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Bacteremia | interventions — Neomycin; Colistin; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neomycin Colistin Nystatin Vancomycin (Experimental): All participating study arm patients will receive SDD from admission to discharge according to the following plan:
  ENTERAL MEDICATION (via feeding tube) x 4 times daily:
  375 mg Neomycin 100 mg Colistin Sulphate
  1 million units Nystatin * 250 mg Vancomycin *
  Nystatin will be prescribed only if there is a positive sputum or urine culture for yeast or candida Vancomycin will be prescribed only in case of a positive screen or culture for MRSA
  Interventions: Drug: Neomycin Colistin Nystatin Vancomycin
- Control (No Intervention): No SDD given for 1 year Screening performed as in intervention arm

INTERVENTIONS:
Drug: Neomycin Colistin Nystatin Vancomycin — All participating study arm patients will receive SDD from admission to discharge
  Other Names: 375 mg Neomycin; 100 mg Colistin Sulphate; 1 million units Nystatin *; 250 mg Vancomycin *
  Arms: Neomycin Colistin Nystatin Vancomycin

SUMMARY:
A simplified graded gut decontamination protocol combined with rigorous bi-weekly screening and appropriate bacterial prophylaxis, will lead to a 25% reduction in the acquisition of blood stream infections and to a 25% reduction in lower airway colonization with multi drug resistant organisms. There will be no concomitant rise in gram-positive or fungal infection or a surgency of new resistance patterns.

DETAILED DESCRIPTION:
Simplified Selective Digestive Tract Decontamination for the prevention of ICU infections in a setting of high-level antibiotic resistance

Scientific Background:

Aerobic gram-negative bacilli (AGNB), Gram-positive bacteria and fungi are responsible for hospital acquired infections. This problem is especially typical in intensive care units (ICUs) due to the complexity of disease and wide use of invasive procedures. The common use of empiric wide-range antibiotic therapy had lead to the development significant resistance of these pathogens and this group of bacteria was defined as Multi-Drug Resistant Organisms (MDRO). Among these bacteria the most important and virulent are: Carbapenem Resistant Enterobacteriaceae (CRE), Extended Spectrum Beta Lactamases (ESBL), Methicillin Resistant Staphylococcus Aureus (MRSA), Vancomycin Resistant Enterococci (VRE) as well as Fluconazol resistant Candida.

The main reservoir of these organisms is the intestinal tract, which raises the possibility that their primary eradication may lead to control of the MDRO epidemic.

Selective Digestive tract Decontamination (SDD) has been studied extensively over the last 10-15 years and there is a body of evidence that shows that this method can reduce acquired infections, bacterial drug resistance and mortality in various ICU settings. It should be pointed out however that many of these studies were performed in units with a low prevalence of infection from MDROs and that they were never performed in units were CREs are endemic. According to the described protocols, SDD was performed as a combination of an a oral antibiotic paste - Selective Oropharyngeal Decontamination (SOD) together with enteral medication given through a gastric feeding tube, as well as a few days of prophylactic intra-venous treatment with an early generation cephalosporin.

This treatment method did not become a standard of care - mostly due to the concern that new resistance will develop to the prescribed enteral antibiotics, or that there will be a rise in the prevalence of other enteral infections as VRE, Clostridium difficile or MRSA acquired infections. Despite evidence that during the SDD treatment period there was actually a reduction of drug resistance, the Center for Disease Control and prevention (CDC) and the protocols of the surviving sepsis campaign do not recommend SDD as a means of coping with the MDRO epidemic. In published SDD protocols there was a use of wide-spectrum antibiotics that covered the range of gram-positive, gram-negative bacteria and fungi, without correlation to the results of primary screening in these patients. Even though this approach did not lead to a rise in bacterial resistance, it raised enough anxiety and resistance within the caregivers to prevent its penetration to daily use. The endemic spread of CRE infection at Rambam Medical Center has lead us to focus on these pathogens in our SDD program, while performing rigorous bi-weekly screening for all bacteria. We gave enteral antibiotic treatment (Neomycin + Polymixin E) targeting AGNB, and only if the primary screening found MRSA or Fungi, did we prescribe enteral preventive treatment against them (Vancomycin or Nystatin). Therefore, a prospective study was performed during 2011 at Rambam department of critical care medicine, on the influence of a simplified SDD protocol on the acquisition of AGNB infection in the ICU. The results show a significant reduction in blood stream infections and a change in the epidemiology of colonization of the respiratory tract - from resistant to sensitive bacteria. There was a concomitant reduction in the use of MDRO- targeted antibiotics.

The proposed multi-center study is based on this successful experience and will focus on the influence of a simplified SDD protocol on colonization and infection with MDROs in israeli ICUs where CREs are endemic.

ELIGIBILITY:
Inclusion Criteria:

1. Expected to be in the ICU > 72 hours
2. Has an enteral feeding tube and can receive enteral medication
3. Has a tracheal tube

Exclusion Criteria:

1. Pt. is moribund - not expected to survive > 28 days
2. Pt. or legal representative refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Number of Intensive care acquired infections per 1000 device days | two years
  A simplified graded SDD protocol combined with rigorous bi-weekly screening and appropriate bacterial prophylaxis, will lead to a reduction in the acquisition of central venous line blood-stream infections and to a reduction in ventilator associated pneumonia. There will be no concomitant rise in gram-positive or fungal infection or a surgency of new resistance patterns.

SECONDARY OUTCOMES:
The effect of SDD on the morbidity and mortality from MDRO on israeli ICU patients. | two years

OTHER OUTCOMES:
The effect of SDD on bacteriological screening of Israeli ICU patients | two years

CONTACTS AND LOCATIONS:
Overall Officials: Yaron P Bar-Lavie, M.D., Study Chair — Rambam Health Care Campus, Haifa, Israel; Mical Paul, Prof., Principal Investigator — Rambam Health Care Campus, Haifa, Israel
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

REFERENCES:
- [Background] de Jonge E, Schultz MJ, Spanjaard L, Bossuyt PM, Vroom MB, Dankert J, Kesecioglu J. Effects of selective decontamination of digestive tract on mortality and acquisition of resistant bacteria in intensive care: a randomised controlled trial. Lancet. 2003 Sep 27;362(9389):1011-6. doi: 10.1016/S0140-6736(03)14409-1. PMID 14522530
- [Background] de Smet AM, Kluytmans JA, Cooper BS, Mascini EM, Benus RF, van der Werf TS, van der Hoeven JG, Pickkers P, Bogaers-Hofman D, van der Meer NJ, Bernards AT, Kuijper EJ, Joore JC, Leverstein-van Hall MA, Bindels AJ, Jansz AR, Wesselink RM, de Jongh BM, Dennesen PJ, van Asselt GJ, te Velde LF, Frenay IH, Kaasjager K, Bosch FH, van Iterson M, Thijsen SF, Kluge GH, Pauw W, de Vries JW, Kaan JA, Arends JP, Aarts LP, Sturm PD, Harinck HI, Voss A, Uijtendaal EV, Blok HE, Thieme Groen ES, Pouw ME, Kalkman CJ, Bonten MJ. Decontamination of the digestive tract and oropharynx in ICU patients. N Engl J Med. 2009 Jan 1;360(1):20-31. doi: 10.1056/NEJMoa0800394. PMID 19118302
- [Background] de Smet AM, Kluytmans JA, Blok HE, Mascini EM, Benus RF, Bernards AT, Kuijper EJ, Leverstein-van Hall MA, Jansz AR, de Jongh BM, van Asselt GJ, Frenay IH, Thijsen SF, Conijn SN, Kaan JA, Arends JP, Sturm PD, Bootsma MC, Bonten MJ. Selective digestive tract decontamination and selective oropharyngeal decontamination and antibiotic resistance in patients in intensive-care units: an open-label, clustered group-randomised, crossover study. Lancet Infect Dis. 2011 May;11(5):372-80. doi: 10.1016/S1473-3099(11)70035-4. Epub 2011 Mar 21. PMID 21420908
- [Background] Schultz MJ, Haas LE. Antibiotics or probiotics as preventive measures against ventilator-associated pneumonia: a literature review. Crit Care. 2011;15(1):R18. doi: 10.1186/cc9963. Epub 2011 Jan 13. PMID 21232110
- [Background] van Saene HK, Petros AJ, Ramsay G, Baxby D. All great truths are iconoclastic: selective decontamination of the digestive tract moves from heresy to level 1 truth. Intensive Care Med. 2003 May;29(5):677-90. doi: 10.1007/s00134-003-1722-2. Epub 2003 Apr 10. PMID 12687326
- [Background] Silvestri L, van Saene HK, Milanese M, Gregori D, Gullo A. Selective decontamination of the digestive tract reduces bacterial bloodstream infection and mortality in critically ill patients. Systematic review of randomized, controlled trials. J Hosp Infect. 2007 Mar;65(3):187-203. doi: 10.1016/j.jhin.2006.10.014. Epub 2007 Jan 22. PMID 17244516